CLINICAL TRIAL: NCT05116956
Title: SKin and Soft Tissue Necrotizing INfections in the Intensive Care Unit: a Prospective Multi-national Cohort Study
Acronym: SKIN-ICU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Henri Mondor University Hospital (Other)
Collaborators: European Society of Intensive Care Medicine (Other)
Responsible Party: Principal Investigator, Nicolas de Prost, Professor Nicolas de Prost, Henri Mondor University Hospital
Other Study IDs: 1-0_30042021
Record Dates: First submitted 2021-10-15; First posted 2021-11-11 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Necrotizing Fasciitis; Fournier Gangrene; Necrotizing Soft Tissue Infection
Keywords: necrotizing soft tissue infection; Necrotizing Fasciitis; Fournier Gangrene
MeSH Terms: conditions — Fasciitis, Necrotizing; Fournier Gangrene

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: non interventional — Multinational prospective, standard care data collection, non-interventional, study not involving human subjects

SUMMARY:
Necrotizing soft-tissue infections (NSTI) are rare and life-threatening bacterial infections characterized by subcutaneous tissue, fascia or muscle necrosis. Few prospective studies have been performed and our current knowledge on NSTI is mostly derived from retrospective single center studies. The "SKin and soft tissue necrotizing INfections in the ICU" (SKIN-ICU) study is a multinational prospective non-interventional cohort study that will include patients admitted to the ICU/intermediate care unit for NSTI or not.

The objectives of the study are :

1. To assess hospital (i.e., ICU and hospital mortality) and medium-term (day-90 mortality, functional outcomes and health-related quality of life scores, HR-QoL) outcomes
2. To report the clinical presentation and microbiological epidemiology of NSTI and identify independent prognostic factors of mortality and altered quality of life

DETAILED DESCRIPTION:
Necrotizing soft-tissue infections (NSTI) are rare and life-threatening bacterial infections characterized by subcutaneous tissue, fascia or muscle necrosis. The mortality of NSTIs is high, ranging from 9% in non-selected patients to up to 30% in the most severe forms requiring intensive care unit (ICU) admission .

With an incidence of 4/100 000 persons per year, initial misdiagnosis is frequent, with no reliable diagnostic test available, frequently leading to a delayed surgical debridement of infected tissues, one of the main modifiable prognostic factors. According to international recommendations, any cutaneous infection associated with the failure of one or more organs or showing a dramatic deterioration must include the diagnosis of NSTI for consideration, even if there is no local sign of the condition being severe. The diagnosis is confirmed by identifying during surgery deficient tissue, sometimes necrotic, which comes away easily in the fingers and by the presence of the typical, foul-smelling "dishwasher" exudate.

The early management of NSTIs is challenging and requires a coordinated and multidisciplinary approach. Treatment of NSTIs consists of early broad-spectrum antimicrobial therapy together with emergency and aggressive surgical debridement including excision of all necrotic and infected tissues. Few prospective studies have been performed and our current knowledge on NSTI is mostly derived from retrospective single center studies.The few randomized therapeutic trials testing interventions in this setting have been disappointing, in part because of the difficulty to identify subgroups for individualized treatments. A large international study aimed at collecting granular data on the clinical presentation, microbiology, management and outcomes of patients with NSTI admitted in the ICU and involving a large number of centers and countries is thus desirable to improve our knowledge on this devastating condition.

The "SKin and soft tissue INfections in the ICU" (SKIN-ICU) study is a multinational prospective non-interventional cohort study that will include patients with NSTI admitted or not to the ICU/intermediate care unit and aim at addressing the following points: 1) Hospital (i.e., ICU and hospital mortality) and medium-term outcomes (three- and six-month survival, functional outcomes and health-related quality of life scores, HR-QoL); and 2) Clinical presentation and microbiological epidemiology of NSTI.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patient with surgically-confirmed NSTI (i.e., macroscopic appearance of tissue during surgery revealing swollen, dull gray tissues with a thin, brownish exudate with or without necrosis)

Exclusion Criteria:

* Patient deprived of liberty by judicial or administrative decision or patient under guardianship
* Expressed opposition to project's participation at the project

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient with surgically-confirmed NSTI
Sampling Method: Probability Sample
Enrollment: 1033 (Estimated)
Dates: Start 2021-11-08 (Actual); Primary Completion 2023-07-22 (Estimated); Study Completion 2023-07-22 (Estimated)

PRIMARY OUTCOMES:
mortality | day 90

SECONDARY OUTCOMES:
Functional outcome | day 90
  Activity of daily living (ADL, 6 questions on selfcare, household, employment, shopping, travel, and communication, each rated 0 (best performance), 1 or 2 (worst performance). An ADL score of 12 indicates a high level of dependence.
Health-related quality of life outcome | day 90
  EuroQol five-dimensional descriptive system (EQ-5D-5L score). It is based on a descriptive system that defines health in terms of 5 dimensions: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression. Each dimension has 3 response categories corresponding to no problems, some problems, and extreme problems. The instrument is designed for self-completion, and respondents also rate their overall health on the day of the interview on a 0-100 hash-marked, vertical visual analogue scale (EQ-VAS).
Microbiology | During the first 72 hours of hospital admission
  Microorganisms involved in blood cultures and per operative tissue samples (species, antibiogram, resistance and "difficult to treat" status)
Skin grafting and amputation | At day 90
  Skin grafting and limb amputation performed within three months of hospital admission will be recorded
SAPS II score | Within 24 hours of hospital admission
  The Simplified Acute Physiology Score II (SAPS II) is a severity of disease score, which is associated with the probability of death at intensive care unit admission (the greater the value of the SAPS II, the greater the odd of death increases).
SOFA score | Within 24 hours of hospital admission
  The Sequential Organ Failure Assessment score is a severity of illness score used in sepsis.the greater the value of the SOFA, the greater the odd of death increases
Anatomic location | Within 24 hours of hospital admission
  Llimbs upper or lower, abdomino-perineal, neck/head, periarticular/circonferential involvement
Body surface area involved | Within 24 hours of hospital admission
  Quantified with the Wallace rule of nine
Portal of entry of the NSTI | Within 24 hours of hospital admission
  Portal of entry of the NSTI will be recorder (e.g., skin ulcer, trauma, other)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas de Prost, MD, PhD, Principal Investigator — Service MIR, Hôpital Henri Mondor
Locations (1):
- Hopital Henri Mondor, Créteil, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stevens DL, Bryant AE. Necrotizing Soft-Tissue Infections. N Engl J Med. 2017 Dec 7;377(23):2253-2265. doi: 10.1056/NEJMra1600673. No abstract available. PMID 29211672
- [Background] Urbina T, Canoui-Poitrine F, Hua C, Layese R, Alves A, Ouedraogo R, Bosc R, Sbidian E, Chosidow O, Dessap AM, de Prost N; Henri Mondor Hospital Necrotizing Fasciitis Group. Long-term quality of life in necrotizing soft-tissue infection survivors: a monocentric prospective cohort study. Ann Intensive Care. 2021 Jul 2;11(1):102. doi: 10.1186/s13613-021-00891-9. PMID 34213694
- [Background] Stevens DL, Bisno AL, Chambers HF, Dellinger EP, Goldstein EJ, Gorbach SL, Hirschmann JV, Kaplan SL, Montoya JG, Wade JC. Practice guidelines for the diagnosis and management of skin and soft tissue infections: 2014 update by the infectious diseases society of America. Clin Infect Dis. 2014 Jul 15;59(2):147-59. doi: 10.1093/cid/ciu296. Epub 2014 Jun 18. PMID 24947530
- [Background] Peetermans M, de Prost N, Eckmann C, Norrby-Teglund A, Skrede S, De Waele JJ. Necrotizing skin and soft-tissue infections in the intensive care unit. Clin Microbiol Infect. 2020 Jan;26(1):8-17. doi: 10.1016/j.cmi.2019.06.031. Epub 2019 Jul 5. PMID 31284035
- [Background] Madsen MB, Skrede S, Bruun T, Arnell P, Rosen A, Nekludov M, Karlsson Y, Bergey F, Saccenti E, Martins Dos Santos VAP, Perner A, Norrby-Teglund A, Hyldegaard O. Necrotizing soft tissue infections - a multicentre, prospective observational study (INFECT): protocol and statistical analysis plan. Acta Anaesthesiol Scand. 2018 Feb;62(2):272-279. doi: 10.1111/aas.13024. Epub 2017 Oct 29. PMID 29082520